CLINICAL TRIAL: NCT03993431
Title: Influence of Luting Cement on the Clinical Outcomes of Zirconia Pediatric Crowns. A 3 Year Split-Mouth Randomized Controlled Trial
Brief Title: Influence of Luting Cement on the Clinical Outcomes of Zirconia Pediatric Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Maha Moussa Azab, Lecturer of Pediatric Dentistry, Faculty of Dentistry, Fayoum University, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zirconia crowns cementation
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Deep Caries
Keywords: Cementation; Zirconia crowns
MeSH Terms: interventions — fuji IX

STUDY DESIGN:
Intervention Model Description: split mouth
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-active cement (Experimental): Bio-active cement dispensed into the crown, and the crown was properly positioned over the tooth, cement was allowed to self-set for 20 seconds while maintaining gentle pressure on the crown, then flash cured using a light curing unit to remove excess cement, buccal and lingual surfaces were light cured for extra 10 seconds each.
  Interventions: Drug: Bio-active cement
- Packable glass ionomer (Active Comparator): Dentin conditioner was applied to the prepared crown surfaces for 20 sec, then rinsed, and dried. Capsule was activated, mixed for 10 seconds in an amalgamator, then loaded into the capsule applier to extrude cement directly into the crown, the crown was properly positioned over the tooth, cement was allowed to self-set for 2 minutes while maintaining gentle pressure on the crown, excess cement was removed before complete setting of cement.
  Interventions: Drug: Packable glass ionomer

INTERVENTIONS:
Drug: Bio-active cement — A cement used for crown cementation, specially recommended for pediatric esthetic crowns
  Other Names: Bio-cem
  Arms: Bio-active cement
Drug: Packable glass ionomer — Glass ionomer cement with improved mechanical properties usually used for restoration of simple small cavities and in Atraumatic Restorative Treatment
  Other Names: Fuji IX; High viscosity glass ionomer
  Arms: Packable glass ionomer

SUMMARY:
The purpose of this split-mouth study was to compare the efficacy of using Bio-active cement versus Packable glass ionomer for cementation of posterior zirconia pediatric crowns.

DETAILED DESCRIPTION:
Restoration of pulp treated or badly broken down deciduous teeth with full coverage restoration have shown superior success rate to all other restorative materials.

Restoration of deciduous teeth with esthetic full coverage restoration has been a challenging aim especially for the more functionally loaded posterior teeth. Due to the continuous increase in socio-economic standards; restoring posterior teeth with esthetic restoration is on high demand nowadays.

The recently introduced zirconia pediatric crowns have been very promising in terms of strength and toughness. Clinical trials on maxillary incisors have shown very high success rates in terms of retention and gingival health.

The problem of restoring posterior deciduous teeth with pre-fabricated zirconia crowns is that its retention is only and totally dependent on luting cement, in addition to the problem of the deteriorated gingival condition around crowns in general.

Being recently introduced to the market; there have not been any clinical trials studying retention of zirconia posterior pediatric crowns published yet.

Recently introduced bio-active cement [NuSmile® BioCem™] is claimed by the manufacturer to be the solution of this problem due to the shock absorbing effect, bioactive components, and antimicrobial effect making it tougher than traditional cements and more gingival friendly.

Also, experienced clinicians have found that packable glass ionomer gives very acceptable results for retention of zirconia pediatric crowns. This may be due to the fact that, pre-fabricated pediatric crown is not well adapted to the prepared tooth creating a greater gap between the prepared tooth and the crown, resulting in a greater film thickness of luting cement, which may benefit from the stronger, tougher and less soluble packable glass ionomer rather than the conventional glass ionomer cement for cementation of zirconia crowns.

There is no clear evidence whether it's better to cement zirconia based crowns with conventional or adhesive cement; and to the investigator's knowledge, there is no data available for the best clinical practice in cementation of zirconia pediatric crowns; and so, this study was carried out to compare the effectiveness of bio-active cement with packable glass ionomer when used for cementation of zirconia pediatric crowns.

ELIGIBILITY:
Inclusion Criteria:

1. 4-7 years old patients having two contra-lateral mandibular first primary molars indicated for restoration with crowns.
2. Presence of sound tooth structure at the cervical margins of the teeth.
3. Presence of opposing functioning teeth.
4. Included teeth should be assessed clinically as free from active pulpal or periodontal conditions.
5. Patient must be in general good health, with no medical contraindication to dental treatment.
6. Patient must be available for required recalls as outlined in the protocol.

Exclusion Criteria:

1. Teeth with defects like hypoplasia or hypocalcification.
2. Patients with untreated periodontal disease.
3. Patients with any pathological or systemic problems that would not allow the dental procedures in this study to take place.
4. Teeth that exhibit mobility.
5. Patients that show signs of severe bruxism or teeth clenching.
6. Subjects with deleterious oral habits like pencil/pen chewing.
7. Uncooperative patients.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of debonded crowns | 1 week
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 1 month
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 3 months
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 6 months
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 9 months
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 12 months
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 18 months
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 24 months
  Binary outcome (debonded/not debonded), assessed by examination
Number of debonded crowns | 36 months
  Binary outcome (debonded/not debonded), assessed by examination

SECONDARY OUTCOMES:
Number of fractured crowns | 1 week, 1, 3, 6, 9, 12, 18, 24 and 36 months
  Binary outcome (Fractured/not fractured), assessed by examination

OTHER OUTCOMES:
Gingival condition | 1 week, 1, 3, 6, 9, 12, 18, 24 and 36 months
  Ordered categorical, assessed by calculating gingival index (0: no inflammation, 1: mild inflammation, 2: moderate inflammation, 3: severe inflammation)

IPD SHARING:
Plan to Share IPD: No